CLINICAL TRIAL: NCT04603794
Title: Comparison of Normal Saline, Hydrogen Peroxide, Chlorhexidine and Povidone-Iodine Mouth Rinses in COVID-19 Patients
Brief Title: Efficacy of Mouthwash in Reducing Salivary Carriage of COVID-19
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, David Hall, Associate Professor, Hospital Attending, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2020H0346
Record Dates: First submitted 2020-10-21; First posted 2020-10-27 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: COVID-19
Keywords: Mouthwashes; COVID-19; Salivary Carriage; Povidone-Iodine; PCR (Polymerase Chain Reaction); Dental Aerosols
MeSH Terms: conditions — COVID-19; Pathologic Complete Response | interventions — Povidone-Iodine; chlorhexidine gluconate; Hydrogen Peroxide; Saline Solution; Fluoridation

STUDY DESIGN:
Intervention Model Description: This randomized, cross-sectional, double blinded, negative controlled, four armed, prospective, interventional study compared Normal Saline, Hydrogen Peroxide, Chlorhexidine and Povidone-Iodine Mouth Rinses in 60 subjects being treated for Covid 19 at the The Ohio State University Medical Center. Real time reverse transcriptase quantitative PCR measured viral loads.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double Blinded. All mouthwash vials are masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- 1% Hydrogen Peroxide Mouth Rinse (Active Comparator): 30 second oral rinse with 1% Hydrogen Peroxide
  Interventions: Drug: 1% Hydrogen Peroxide
- 0.12% Chlorhexidine Gluconate Mouth Rinse (Active Comparator): 30 second oral rinse with 0.12% Chlorhexidine Gluconate
  Interventions: Drug: 0.12% Chlorhexidine Gluconate Mouth Rinse
- 0.5% Povidone Iodine Mouth Rinse (Active Comparator): 30 second oral rinse with 0.5% Povidone Iodine Mouth wash
  Interventions: Drug: 0.5% Povidone Iodine
- 0.9% Normal Saline Mouth Rinse (Placebo Comparator): 30 second oral rinse with 0.9% Normal Saline
  Interventions: Drug: 0.9% Normal Saline

INTERVENTIONS:
Drug: 0.5% Povidone Iodine — Commercially Available Mouth Rinses and Over the Counter Standard Formulations
  Other Names: Betadine Mouthwash
  Arms: 0.5% Povidone Iodine Mouth Rinse
Drug: 0.12% Chlorhexidine Gluconate Mouth Rinse — Commercially Available Mouth Rinses
  Other Names: Peridex
  Arms: 0.12% Chlorhexidine Gluconate Mouth Rinse
Drug: 1% Hydrogen Peroxide — Commercially Available Over the Counter Standard Formulations USP (United States Pharmacopeia)
  Other Names: Hydrogen Peroxide
  Arms: 1% Hydrogen Peroxide Mouth Rinse
Drug: 0.9% Normal Saline — Commercially Available Over the Counter Standard Formulations USP (United States Pharmacopeia)
  Other Names: Salt Water
  Arms: 0.9% Normal Saline Mouth Rinse

SUMMARY:
Researchers know that the virus that causes COVID-19 has been found in the saliva (spit) of individuals who exhibit signs of the disease. Investigators would like to test the ability of three mouthwashes to reduce the levels of this virus in participants' mouths. Investigators will ask participants to use a liquid to swish around in the mouth for 30 seconds and spit it into a collection cup. Investigators will also collect spit from participants before and after participants use the mouthwash. Although participants will have no direct benefits from the study, investigators will gain a wealth of information that would benefit patients who are at risk for COVID-19.

DETAILED DESCRIPTION:
Project aims:

Aim 1: To examine the salivary carriage of COVID-19 in individuals before and after use of mouthwashes known to reduce oral microbiota, using real time reverse transcriptase quantitative PCR (Polymerase Chain Reaction) to quantify viral load.

RESEARCH STRATEGY:

A. Recruitment and baseline data:

This is a cross-sectional interventional 4 arm study. 60 subjects between 18-80 years of age will be recruited from those who are being treated for COVID-19 at the Ohio State University Medical Center. There is no data upon which to base sample size estimates, and investigators have landed on this number in an effort to obtain a representative sample of Ohio's population. If the potential subject is interested in participating, the study coordinator will collect contact information from the candidate and the consent form will be presented to these individuals. Subjects will be allowed sufficient time to read and ask questions, and once sign these forms, a detailed history including information about ethnicity, education, income, age, sex, race, medical status (including pregnancy) and dental history will be elicited. Subjects will self-collect saliva in a 5 ml collection tube, following which they will be asked to use one of 3 mouthwashes (chlorhexidine, povidone iodine, hydrogen peroxide or control(saline) for thirty seconds and spit them into collection tubes. Investigators will use Peridex, Hydrogen Peroxide and Betadine, which are commercially available formulations of chlorhexidine, hydrogen peroxide and betadine respectively, to reduce formulation bias. Investigators have attached the product labels as appendices to this proposal. The exact mouthwash will be decided by random chance using a random number generator. Investigators have generated the following randomization schedule using Microsoft excel: Each subject will be assigned a number as they are recruited (E.g. first patient to sign the consent will be patient 1, and the second will be patient 2 and so on). Patients 1 and 2 will receive saline and 3 will receive chlorhexidine etc. base on the above randomization schedule. Subjects will then collect saliva in separate collection tubes 15 and 30 minutes after rinsing.

B. Sample collection Saliva will be collected using a methodology described by previous investigators. Briefly, subjects will be asked to collect saliva in their mouth for 3 minutes and then continuously drool into a tube for 3 minutes. This method will allow investigators to collect unstimulated saliva. Saliva will be collected using kits containing RNA (Ribonucleic Acid) stabilizer (Oragen RNA kit).

C. Measurement / Instrumentation

Total RNA will be isolated from saliva using the mirVana miRNA (Messenger Ribonucleic Acid) isolation kit (Applied Biosystems). Microbial cells will be lysed and RNA will be extracted by Acid-Phenol:Chloroform and ethanol precipitation and eluted in nuclease-free water. Investigators will use well validated primers to quantify copy numbers of COVID-19 spike protein mRNA (Messenger Ribonucleic Acid) from the saliva. For an absolute quantification of COVID-19, investigators will use one step RT-PCR (Reverse Transcriptase) assay by using an appropriate commercially available kit. In this step investigators will convert mRNA to cDNA (complementary Deoxyribonucleic Acid) and then quantify the cDNA by using targeted primers and then copy numbers of the COVID-19 will be calculated by comparing ct (cycle threshold)Values samples against standard curve. In order to generate standard curves for absolute quantification, target genes will be amplified with PCR. The PCR products will be cloned into suitable vector. Then plasmids will be extracted, serially diluted, and used as templates in qPCR (quantitative polymerase chain reaction) for generating standard curves.

D. Internal Validity Subjects will be recruited randomly through voluntary participation. This will eliminate presentation bias.

E. Data Analysis

Descriptive statistics will be provided as estimates of salivary carriage of COVID-19. Frequency of salivary carriage of the virus will be expressed as a percent of the total sample population. Reduction in COVID-19 following mouthwash use will be expressed as fold change and compared between the three mouthwash groups using parametric tests.

ELIGIBILITY:
Inclusion Criteria:

1. adults age 18-80 admitted to The Ohio State University Medical Center,
2. diagnosis of COVID-19 confirmed by Polymerase Chain Reaction (PCR),
3. salivary carriage of COVID-19 virus
4. ability to perform mouthwash rinses and to expectorate.

Exclusion Criteria:

1. allergy to any study mouth rinse,
2. active uncontrolled thyroid disease,
3. pregnancy
4. patients undergoing radioactive iodine therapy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2020-11 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
real time reverse transcriptase quantitative PCR | 3 measurements of changes from times 0 minutes. vs:15 minutes, and vs: 45 minutes during a single session
  Saliva load was expressed in copies x 10 8 of COVID-19 RNA
ct values | 3 measurements of changes from times 0 minutes.vs:15 minutes, and vs:45 minutes during a single session
  cycle thresholds

CONTACTS AND LOCATIONS:
Overall Officials: David L Hall, DDS, Study Director — The Ohio State University College of Dentistry
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
As per The Ohio State University Office for Responsible Research Practices (Human Studies IRB)

REFERENCES:
- [Background] Serban D, Banu A, Serban C, Tuta-Sas I, Vlaicu B. Predictors of quantitative microbiological analysis of spatter and aerosolization during scaling. Rev Med Chir Soc Med Nat Iasi. 2013 Apr-Jun;117(2):503-8. PMID 24340537
- [Background] Gupta G, Mitra D, Ashok KP, Gupta A, Soni S, Ahmed S, Arya A. Efficacy of preprocedural mouth rinsing in reducing aerosol contamination produced by ultrasonic scaler: a pilot study. J Periodontol. 2014 Apr;85(4):562-8. doi: 10.1902/jop.2013.120616. Epub 2013 Jul 15. PMID 23855840
- [Background] Shetty SK, Sharath K, Shenoy S, Sreekumar C, Shetty RN, Biju T. Compare the effcacy of two commercially available mouthrinses in reducing viable bacterial count in dental aerosol produced during ultrasonic scaling when used as a preprocedural rinse. J Contemp Dent Pract. 2013 Sep 1;14(5):848-51. doi: 10.5005/jp-journals-10024-1414. PMID 24685786
- [Background] Devker NR, Mohitey J, Vibhute A, Chouhan VS, Chavan P, Malagi S, Joseph R. A study to evaluate and compare the efficacy of preprocedural mouthrinsing and high volume evacuator attachment alone and in combination in reducing the amount of viable aerosols produced during ultrasonic scaling procedure. J Contemp Dent Pract. 2012 Sep 1;13(5):681-9. doi: 10.5005/jp-journals-10024-1209. PMID 23250175
- [Background] Klyn SL, Cummings DE, Richardson BW, Davis RD. Reduction of bacteria-containing spray produced during ultrasonic scaling. Gen Dent. 2001 Nov-Dec;49(6):648-52. PMID 12024755
- [Background] Wirthlin MR, Choi JH, Kye SB. Use of chlorine dioxide mouthrinse as the ultrasonic scaling lavage reduces the viable bacteria in the generated aerosols. J West Soc Periodontol Periodontal Abstr. 2006;54(2):35-44. No abstract available. PMID 17214015
- [Background] Peng X, Xu X, Li Y, Cheng L, Zhou X, Ren B. Transmission routes of 2019-nCoV and controls in dental practice. Int J Oral Sci. 2020 Mar 3;12(1):9. doi: 10.1038/s41368-020-0075-9. PMID 32127517
- [Background] Navazesh M. Methods for collecting saliva. Ann N Y Acad Sci. 1993 Sep 20;694:72-7. doi: 10.1111/j.1749-6632.1993.tb18343.x. No abstract available. PMID 8215087
- [Background] To KK, Tsang OT, Yip CC, Chan KH, Wu TC, Chan JM, Leung WS, Chik TS, Choi CY, Kandamby DH, Lung DC, Tam AR, Poon RW, Fung AY, Hung IF, Cheng VC, Chan JF, Yuen KY. Consistent Detection of 2019 Novel Coronavirus in Saliva. Clin Infect Dis. 2020 Jul 28;71(15):841-843. doi: 10.1093/cid/ciaa149. PMID 32047895
- [Derived] Chaudhary P, Melkonyan A, Meethil A, Saraswat S, Hall DL, Cottle J, Wenzel M, Ayouty N, Bense S, Casanova F, Chaney M, Chase H, Hermel R, McClement M, Sesson C, Woolsey B, Kumar P. Estimating salivary carriage of severe acute respiratory syndrome coronavirus 2 in nonsymptomatic people and efficacy of mouthrinse in reducing viral load: A randomized controlled trial. J Am Dent Assoc. 2021 Nov;152(11):903-908. doi: 10.1016/j.adaj.2021.05.021. Epub 2021 Jun 11. PMID 34561086
- See also: Povidone-iodine demonstrates rapid in-vitro Activity... — https://doi.org/10.21203/rs.3.rs-34544/v2
- See also: Viral dynamics in asymptomatic patients with COVID-19 — https://doi.org/10.1016/j.ijid.2020.05.030